CLINICAL TRIAL: NCT01961570
Title: Clinical Evaluation of the Articulinx InterCarpoMetacarpal Cushion (ICMC) for Osteoarthritis of the First CarpoMetacarpal Joint: A New Study of the ICMC in a Clinical Setting
Brief Title: Clinical Evaluation of the Articulinx InterCarpoMetacarpal Cushion (ICMC)for Osteoarthritis of the First CarpoMetacarpal Joint
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Articulinx (Industry)
Responsible Party: Sponsor
Other Study IDs: CL 0031
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Early Stage Osteoarthritis of the CMC-1 Joint
Keywords: Early stage hand osteoarthritis; Carpometacarpal osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to evaluate the performance of the Articulinx ICMC (InterCarpoMetacarpalCushion)in the carpometacarpal joint (CMC joint) and to describe the clinical results in patients who have been treated with this device. Expected results include the relief of symptoms and improvement of function in patients with symptomatic osteoarthritis (OA) of the CMC-1 joint. Evaluation of device performance will be achieved through measurements of pain, pain medication use, and joint function in up to 20 subjects. Each subject will be compared to their pre-surgery status for each endpoint.

DETAILED DESCRIPTION:
The Articulinx ICMC is a minimally invasive orthopedic device intended to be implanted into the basilar, or first carpometacarpal (CMC) joint, as an interpositional spacer between the first metacarpal and trapezium bones. The device is intended to be used in the treatment of thumb disabilities resulting from osteoarthritis of the CMC-1 joint.

The Articulinx ICMC is a molded polymer disc with an encapsulated radiopaque marker. The Articulinx ICMC is designed to be an inter-positional spacer for the treatment of symptoms of early-stage osteoarthritis of the first CMC joint. When properly positioned in the joint, the ICMC can preserve or restore normal space between the trapezium and thumb metacarpal bones in the first CMC joint. The restoration of natural spacing and biomechanics within the joint is expected to reduce pain and restore strength and function.

The ICMC is designed to be implanted earlier in the OA disease process than other basilar joint implants. The ICMC allows a more active lifestyle and may reduce or eliminate the need for long-term use of prescribed arthritis medications. Because the ICMC procedure does not remove supportive bone or tissue, the procedure is reversible and treatment options for later stage disease progression remain available to patients.

The ICMC was first placed on the EU (European Union) market by the Sponsor in April, 2011 following approval to carry the CE (European Community) Mark based upon successful pre-clinical and clinical testing. In other clinical studies, one single site study and one multicenter site study, both conducted in accordance with ISO 14155 (International Standards Organization), the 1-year enrollment is completed and 2-year follow-up is ongoing.

The primary objective of this study is to document the safety of the Articulinx ICMC by evaluating Incidence of unanticipated device and procedure related adverse events intra-operatively, and through one year follow-up.

The secondary objectives of this study are to describe clinical and radiographic outcomes in patients who are treated with the device.

This is a single site study in The Netherlands. Study enrollment will begin following required regulatory submissions/Ethics Committee approval and after site study personnel training is completed. The study will be conducted in conformance with ISO 14155 and will evaluate the performance of the Articulinx ICMC for the relief of the symptoms of osteoarthritis in the CMC-1 joint. Primary and secondary study endpoints will be evaluated through one year and patients will continue to be followed for two years for evaluation of longer-term performance.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed by the investigator to be medically acceptable for a surgical procedure?
* Patient is aged 40 to 75 inclusive?
* Patient has symptomatic osteoarthritis of the carpometacarpal (CMC-1) joint as demonstrated by a minimum DASH score of 40 at baseline?
* Patient has pain in the target CMC joint as demonstrated by an average VAS pain score greater than or equal to 40 at baseline on a 100mm VAS?
* Patient has radiographic evidence of Stage II OA with no free-floating bodies in the CMC-1 joint?
* Radiographic Stage II OA is defined according to the Eaton-Glickel classification system (based upon lateral view) as follows:

"Slight narrowing of the TM [trapezio-metacarpal/CMC] joint will be present with minimal sclerotic changes of the subchondral bone. There may be joint debris not exceeding 2 mm in diameter in the form of osteophytes or loose bodies The ST [scapho-trapzeial joint] should appear normal."

* Patient has subluxation of less than one-third of the target CMC joint?
* Patient agrees to return to the clinic for follow-up visits at the required times per protocol and follow the requirements of this protocol?
* Patient is able and willing to provide voluntary consent to participate?

Exclusion Criteria:

* Patient has non-symptomatic osteoarthritis of the first CMC joint?
* Patient has small bone or calcific fragments (spurs, osteophytes) in the target CMC joint greater than two millimeters (>2mm) in diameter?
* Patient has free floating bodies of any size within the target CMC joint?
* Patient has radiographic/imaging evidence of significant osteoarthritic changes within the first metacarpal, or scaphotrapezotrapezoidal (STT) joint of the target wrist consistent with Stage III/IV OA, according to Eaton-Glickel, as defined below?

"Stage III OA: The joint space will be markedly narrowed or obliterated with cystic changes, sclerotic bone, varying degrees of dorsal subluxation, and joint debris exceeding 2 mm in diameter. The ST joint will appear normal."

"Stage IV OA: There is complete deterioration of the TM [CMC] joint as in stage III and, in addition, the ST joint will be narrowed with sclerotic and cystic changes apparent."

* Patient has concomitant musculoskeletal pathology of the target hand, such as carpal tunnel syndrome, palmar tenosynovitis, scaphoulnate ligament instability/degeneration, ulnocarpal impaction syndrome, or trigger finger;
* Patient has concomitant rheumatic disease (e.g., inflammatory rheumatoid arthritis, cutaneous psoriasis, polyarticular chondrocalcinosis, gout, fibromyalgia) or exhibits signs of metabolic disorders affecting the bone or joint (e.g., osteoporosis, osteomalacia, hyper- or hypo-parathyroidism, Paget's disease)?
* Patient has an active infection, sepsis or osteomyelitis?
* Patient has skin disease or eruption at the CMC target site?
* Patient had previous surgery on the target CMC joint or on the wrist of the target hand?
* Patient had significant injury to the target CMC joint within the 6 months prior to study enrollment or a significant permanent injury at any time prior to study enrollment?
* Patient has a significant comorbid medical condition that could exacerbate pain symptoms or adversely affect physical functioning or healing of the thumb CMC joint (e.g. de Quervains disease, Ehlers-Danlos Syndrome, Complex Regional Pain Syndrome)?
* Patient has had corticosteroid injections in the target CMC joint within 6 months prior to study enrollment?
* Patient takes concomitant immunosuppressive therapy (e.g., oral/injectable glucocorticoids, alkylating agents, antimetabolites, antibodies, drugs acting on immunophilins [Ciclosporin, Sirolimus], interferons, opioids) that could adversely affect healing?
* Patient has uncontrolled diabetes mellitus?
* Patient takes anticoagulation and or antiplatelet therapy that cannot be stopped prior to surgery?
* Patient is planning a pregnancy, or patient is pregnant and/or lactating? (If a subject becomes pregnant after enrollment in the study, then the subject will continue to be followed, even though she may miss some follow-up appointments. During the pregnancy, X-rays will not be performed.)
* Patient is participating in any other clinical investigation that could impact the outcome of this study?
* Patient has a known history of drug or alcohol abuse in the previous 12 months?
* Patient has a history of, or is currently engaged in, litigation for musculoskeletal injuries or disorders or medical malpractice?
* Patient has other life circumstances that the Investigator feels would interfere with study participation such as planned relocation, difficulty complying with schedule of study follow-up visits, is generally uncooperative?

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women with early stage carpometacarpal-1 (CMC-1)joint osteoarthrititis.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study is the Incidence of unanticipated device and procedure related adverse events. | Intra-operatively and through one year follow-up.
  Reported incidence of unanticipated device and procedure related Adverse Events will be documented at all scheduled visits and within 24 hours of knowledge of an event.

SECONDARY OUTCOMES:
Secondary outcome measures describe clinical and radiographic outcomes in patients treated with the device. | Post operative follow-up at 3mo, 6mo, and 12mo
  Changes in CMC-1 joint function post-procedure compared to preoperative baseline
Secondary outcome measures describe clinical and radiographic outcomes in patients treated with the device. | Post operative follow-up at 3mo, 6mo, and 12mo
  Changes in average CMC-1 joint pain score at the one-year postoperative follow-up compared to preoperative baseline
Secondary outcome measures describe clinical and radiographic outcomes in patients treated with the device. | Post operative follow-up at 3mo, 6mo, and 12mo.
  Change in DASH scores post-procedure as compared to preoperative baseline
Secondary outcome measures describe clinical and radiographic outcomes in patients treated with the device. | Postoperative follow-up at 3mo, 6mo, and 12mo
  Maintenance of trapezial joint space height compared to pre-operative baseline

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Marco J.P.F. Ritt, MD, PhD, Principal Investigator — Vrij University (VU) Medical Center
Locations (1):
- Vrij University Medical Center (VUmc), Amsterdam, Netherlands